CLINICAL TRIAL: NCT00197873
Title: Randomized, Double Blind, Placebo Controlled, Cross-over Phase II Study on the Effects of Lactobacillus Rhamnosus GG Supplementation in Patients on 1st Line XELOXA Treatment for Metastatic Colorectal Cancer
Brief Title: Lactobacillus Rhamnosus in Prevention of Chemotherapy-related Diarrhoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Heikki Joensuu, professor, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ML18581
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; probiotics; chemotherapy; prevention; adverse effects; diarrhoea
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactophilus (Active Comparator): Lactophilus supplementation
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus supplementation
- Placebo (Placebo Comparator): Placebo is administered during chemotherapy.
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus supplementation; Other: Placebo administration.

INTERVENTIONS:
Dietary Supplement: Lactobacillus Rhamnosus supplementation — Lactophilus supplementation is administered during chemotherapy.
  Other Names: Probiotics
Other: Placebo administration. — Placebo is administered during chemotherapy.
  Other Names: Placebo.
  Arms: Placebo

SUMMARY:
Chemotherapy may cause diarrhoea, which may be associated with treatment delay and infections. The purpose of the study is to investigate whether oral supplementation with lactobacilli will alleviate chemotherapy related diarrhoea. Patients diagnosed with advanced colorectal cancer and who will receive chemotherapy will be randomly assigned to receive either lactobacilli or placebo during chemotherapy. The study is a prospective, multicenter, randomized, double-blind, placebo-controlled study. The primary outcome measure is frequency of moderate/severe diarrhoea. The study will also address safety and tolerability of chemotherapy, response to chemotherapy, and serum growth factor levels.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, cross-over, double-blind, placebo-controlled study. Patients diagnosed with advanced colorectal cancer with overt distant metastases and who will receive chemotherapy consisting of capecitabine, oxaliplatin and bevacizumab, given as 3-weekly cycles, will be randomly assigned to receive either lactobacilli (GefilusR) or placebo during the first 3 cycles of chemotherapy (for 9 weeks). Following this, the groups will be crossed over and those study participants who were allocated to lactobacilli will receive placebo for 9 weeks, and vice versa. Lactobacilli and placebo are administered twice daily. The total daily dose of lactobacilli is 20 billion CFU. The primary outcome measure is frequency of moderate/severe diarrhoea (grade 2-4). Adverse effects (including the frequency of diarrhoea, flatulence, bloating, constipation, and nausea) will be longitudinally monitored based on a patient diary and study visits. The study will also address safety and tolerability of chemotherapy, response to chemotherapy, progression-free survival, resectability of liver metastases, and serum growth factor levels. A total of 84 patients are planned to be entered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of CRC, chemotherapy naïve for metastatic disease (prior adjuvant chemotherapy for CRC allowed), who are scheduled to start capecitabine treatment as first line chemotherapy for metastatic disease
* Age 18 or older
* Measurable or non-measurable metastatic disease
* Performance status ECOG performance status 0-2
* Life expectancy greater than 3 months
* Thrombocytes 100,000/µL or greater, neutrophils 1.500/µl or greater, Aspartate amino transferase/Alanine amino transferase <= 2.5 x Upper limit of normal (ULN) (< 5 x ULN if liver metastases present), Alkaline phosphatase <=2.5 x ULN (< 5 x ULN if liver metastases present), Serum bilirubin <= 1.5 x ULN, Serum Creatinine <= 1.5 x ULN, Urine dipstick of proteinuria <2+ (or U-Prot <100mg/dl). Patients discovered to have 2+ or greater proteinuria on dipstick urinalysis at baseline, must undergo a 24-hour urine collection and must have <= 1 g of protein/24 hr
* Women of childbearing potential must have a negative serum pregnancy test done prior to the administration of bevacizumab. Patient and their partner should prevent pregnancy (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) up to at least 6 months after last treatment completion or the last drug dose, whatever happens first
* Signed written informed consent according to ICH/GCP and the local regulations (approved by the Independent Ethics Committee [IEC]) will be obtained prior to any study specific screening procedures
* Patient must be able to comply with the protocol

Exclusion Criteria:

* Prior treatment with first-line chemotherapy for metastatic CRC
* Adjuvant treatment with bevacizumab within 12 months
* Acute or chronic diarrhea or colostomy
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 0 (Patients must have recovered from any major surgery)
* Near future planned radiotherapy for underlying disease (prior completed radiotherapy treatment allowed)
* Clinical or radiological evidence of CNS metastases
* Past or current history within the last 5 years of malignancies except for the indication under this study and curatively treated Basal and squamous cell carcinoma of the skin or In-situ carcinoma of the cervix
* Serious non-healing wound or ulcer
* Evidence of bleeding diathesis or coagulopathy
* Uncontrolled hypertension
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤ 6 months), myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Treatment with any investigational drug (including IMMP, EGFR inhibitors) or participation in another investigational study within 30 days prior to enrolment
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the treatment or patient at high risk from treatment complications
* Ongoing treatment with aspirin (> 325 mg/day), continuous high dose NSAIDS or other medications known to predispose to gastrointestinal ulceration
* Pregnancy (positive serum pregnancy test) and lactation
* Any other serious or uncontrolled illness which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-09; Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Effect on the treatment-related grade 2 to 4 diarrhoea | 18 weeks
  Numbers of bowel movements per day.

SECONDARY OUTCOMES:
Effect on treatment related toxicity other than diarrhea | 18 weeks
  Adverse effects detected in the study groups.
Association between supplementation and response | 18 weeks
  Response rate assessed with imaging.
Effect on resectability of liver metastases | 1 year
  Numbers of liver resections carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, M.D., Study Director — Department of Oncology, Helsinki University Central Hospital
Locations (1):
- Department of Oncology, Helsinki, Finland